CLINICAL TRIAL: NCT05785312
Title: Development of Online EMDR Therapy System and Its Comparative Testing With Face-to-Face EMDR Therapy for Treatment of Anxiety and Depressive Disorders in Pakistan: A Randomized Controlled Feasibility-Pilot Study*
Brief Title: Development of Online EMDR Therapy System and Its Comparative Testing With Face-to-Face EMDR Therapy for Treatment of Anxiety and Depressive Disorders in Pakistan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khushal Khan Khattak Univeristy, Karak, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Anwar Khan, Dr. Anwar Khan, Director and Principal Investigator, Office of Research, Innovation and Commercialization, Khushal Khan Khattak Univeristy, Karak, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12321
Record Dates: First submitted 2023-02-01; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Generalized Anxiety Disorder; Major Depressive Disorder; Social Anxiety Disorder; Somatic Symptom; Panic Attacks; Obsessive-Compulsive Disorder and Symptoms
Keywords: EMDR; Online EMDR; Depression; Anxiety; Pakistan; Pilot Study
MeSH Terms: conditions — Generalized Anxiety Disorder; Depressive Disorder, Major; Phobia, Social; Medically Unexplained Symptoms; Panic Disorder; Obsessive-Compulsive Disorder; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Since this a comparative study, therefore after recruiting patients, the patients will be randomly allocated parallelly to the two arms. Arm One will will be Face-to-Face EMDR Therapy, in which the patients will receive standard EMDR therapy in a face-to-face meeting with the therapist. Arm two will be the online EMDR Therapy, in which the patients will receive EMDR therapy online via video conferencing. The patient will be randomly selected assigned to each arm with 1:1 allocation.
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face to Face Eye Movement Desensitization & Reprocessing Therapy (Experimental): The standard Face to Face Eye Movement Desensitization & Reprocessing Therapy will be applied by a trained clinical psychologist through in person face to face sessions.
  Interventions: Other: Face to Face Eye Movement Desensitization & Reprocessing Therapy
- Online Eye Movement Desensitization & Reprocessing Therapy (Active Comparator): The Online Eye Movement Desensitization & Reprocessing Therapy will be applied by a trained clinical psychologist through computer system by connecting through internet. For this purpose the online EMDR therapy application software will be installed
  Interventions: Device: Online EMDR Therapy System

INTERVENTIONS:
Device: Online EMDR Therapy System — Online EMDR Therapy System will be delivered through online computer system that will be specifically designed for delivering EMDR therapy online
  Arms: Online Eye Movement Desensitization & Reprocessing Therapy
Other: Face to Face Eye Movement Desensitization & Reprocessing Therapy — The Face to Face Eye Movement Desensitization & Reprocessing Therapy will be delivered in person inside clinician's room by following standard EMDR therapy protocol
  Arms: Face to Face Eye Movement Desensitization & Reprocessing Therapy

SUMMARY:
This study aims at developing an online system for the remote delivery of EMDR therapy in Pakistan. Moreover, this study will compare the efficacy of online EMDR therapy with face-to-face EMDR therapy.

DETAILED DESCRIPTION:
Depressive and Anxiety disorders have higher global prevalence. Moreover, they are leading causes of global burden of mental diseases (i.e., 24th leading cause of global Disability-adjusted Life Years). Such increase in the global prevalence of Depression and Anxiety disorders is due to the complexities of modern life. Nowadays various evidence-based psychotherapies, like e.g., EMDR therapy are available. Therapists have been using face-to-face modes for a long time, but with the expansion of Computer Technologies, online psychotherapies have been developed. The need for online psychotherapies was further increased due to Corona Virus-19 pandemic. Scientists have developed online modes of Cognitive Behavioral Therapy, Prolonged Exposure Therapy and Mindfulness Therapy, etc., but there are limited research studies on the online EMDR therapy, especially in the Asian countries. Therefore, questions arises a) Is it possible to treat Anxiety & Depressive disorders through online EMDR therapy? b) What adaptations would be required to be made in the face-to-face protocols of EMDR therapy? c) Whether the online EMDR therapy will be: i) fit and safe for use; ii) usable; iii) operable & practicable; and iv) efficient in delivering a timely treatment? The existing online programs of EMDR Therapy, e.g., VirtualEMDR have been built in the western-developed countries, hence may not be accessible to the local patients in Pakistan. Moreover, these programs might not be compatible with the requirements of patients in Pakistan. Keeping in view such facts, this study aims at developing an online system for the remote delivery of EMDR therapy in Pakistan. Moreover, this study will compare the efficacy of online EMDR therapy with face-to-face EMDR therapy. For this purpose, patients will be recruited through a consecutive sampling technique, with a sample size of n=30. Data on symptomology and other technical data will be collected through standard scales. Qualitative data were analyzed by qualitative techniques, while the quantitative data were analyzed by descriptive and multivariate statistics. This study will be unique in its nature since a) an online EMDR therapy will be developed for Pakistani patients, b) this online system will be scientifically validated, c) and its efficacy will be compared with face-to-face EMDR therapy. This study will provide a base for the future researchers to design and implement online psychotherapies in Pakistan. In this way, the mental healthcare system of Pakistan could be ultimately revolutionized through the online treatment facilities.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients.
2. Patients between the age of 18 to 50 years (since this study is neither on children nor on old patients).
3. Patients who have basic knowledge & skills of computer, mobile and internet (although the recruited patients will be given training for using the online EMDR).
4. Patients do not suffer from severe neuropsychological and cognitive impairments.
5. Patients have not received any pharmacological therapy in the last three months.
6. Patients have not received any other psychotherapy like Cognitive Behavioral Therapy.

Ages: 18 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — both males and females within the age range of 18 to 50 years
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Assessing changes in symptom of Generalized Anxiety Disorder with time (i.e., treatment course) | A total of 40 patients will be selected. Symptoms will be screened for 06 months in such a way that symptoms will be assessed first during base line (T1), then during mid of treatment (T2), and finally at the end of treatment (T3)
  Generalized Anxiety Disorder by Generalized Anxiety Disorder Questionnaire-IV. Score of 5.7 or above will indicate that the patient is suffering from Generalized Anxiety Disorder.
Assessing changes in symptom of Major Depressive Disorder with time (i.e., treatment course) | A total of 40 patients will be selected. Symptoms will be screened for 06 months in such a way that symptoms will be assessed first during base line (T1), then during mid of treatment (T2), and finally at the end of treatment (T3)
  Major Depressive Disorder by Beck Depression Inventory-II. Score of 30 or above will indicate that the patient is suffering from major depressive disorder
Assessing changes in symptom of Social Anxiety Disorder with time (i.e., treatment course) | A total of 40 patients will be selected. Symptoms will be screened for 06 months in such a way that symptoms will be assessed first during base line (T1), then during mid of treatment (T2), and finally at the end of treatment (T3)
  Social Anxiety Disorder will be assed by Social Anxiety Scale. Score of 60 or above will indicate that the patient is suffering from Social Anxiety Disorder.

SECONDARY OUTCOMES:
Assessing changes in Panic symptoms with time (i.e., treatment course) | A total of 40 patients will be selected. Symptoms will be screened for 06 months in such a way that symptoms will be assessed first during base line (T1), then during mid of treatment (T2), and finally at the end of treatment (T3)
  Panic Attacks by Panic Disorder Severity Scale. Score of 20 or above will indicate that the patient is suffering form panic symptoms.
Assessing changes in Somatic symptoms | A total of 40 patients will be selected. Symptoms will be screened for 06 months in such a way that symptoms will be assessed first during base line (T1), then during mid of treatment (T2), and finally at the end of treatment (T3)
  Somatic Symptoms by the Somatic Symptom Scale-8. Score of 11 or above will indicate that the patient is suffering from somatic symptoms.
Assessing changes in Obsessive symptoms with time (i.e., treatment course) | A total of 40 patients will be selected. Symptoms will be screened for 06 months in such a way that symptoms will be assessed first during base line (T1), then during mid of treatment (T2), and finally at the end of treatment (T3)
  Obsessive Compulsive Symptoms by Dimensional Obsessive-Compulsive Scale. Score of 15 or above on each dimension will indicate that the patient is having Obsessive Compulsive Symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kushal Khan University, Lakki, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
will only be shared after placing valid request